CLINICAL TRIAL: NCT02385669
Title: A Phase I/II Trial to Evaluate the Safety and Immunogenicity of a Helper Peptide Vaccine Plus CTLA-4 Blockade in Melanoma Patients (Mel62; 6PAC)
Brief Title: A Phase I/II Trial to Evaluate a Peptide Vaccine Plus Ipilimumab in Patients With Melanoma
Acronym: Mel62; 6PAC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: why study stopped
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17780
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Melanoma
Keywords: vaccine; peptide; ipilimumab; Yervoy; Montanide ISA-51
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 6MHP and ipilimumab (Experimental): The vaccine drug product, 6MHP, consists of 6 class II MHC-restricted peptides derived from melanoma proteins. Each vaccine consists of 200 mcg of each of the six peptides. An aqueous solution of vaccine is mixed 1/1 with Montanide ISA-51 to form water-in-oil emulsions. Vaccines are administered days 1, 8, 15, 43, 64, and 85. All peptide vaccines are administered intradermally and subcutaneously.
  Ipilimumab will be administered in accord with the official prescribing information: 3 mg/kg intravenously once every 3 weeks, for 4 doses. Ipilimumab will be administered on days 1, 22, 43, and 64.
  Interventions: Drug: Ipilimumab; Biological: 6MHP

INTERVENTIONS:
Drug: Ipilimumab — Checkpoint blockade inhibitor
  Other Names: Yervoy
Biological: 6MHP — 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Other Names: 6 melanoma helper peptide vaccine

SUMMARY:
This study evaluates whether it is safe to administer a peptide vaccine with ipilimumab. This study will also evaluate the effects of the combination of the peptide vaccine and ipilimumab on the immune system. The investigators will monitor these effects by performing tests in the laboratory on participants' blood, a lymph node, and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stage IIA (with class 2 DecisionDx Score) through IV melanoma in cohorts defined below. These participants may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. The diagnosis of melanoma must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on the revised AJCC staging system. Participants must be eligible to be treated with ipilimumab based on clinician judgment within standard of care.

  * Cohort 1 (Advanced Patients): unresectable stage III or IV melanoma that have clinical or radiographic evidence of disease.
  * Cohort 2 (Neoadjuvant therapy): primary melanoma with clinically apparent lymph node or in transit/satellite lesions with or without lymph node involvement, in transit recurrence or metastatic recurrence amenable to complete resection to no evidence of disease
  * Cohort 3 (Adjuvant therapy): Stage IIA (with class 2 DecisionDx Score), IIB-IV melanoma resected to no evidence of disease.
* Participants will be required to have radiological studies to define radiologically evident disease. Required studies include:

  * Chest CT scan,
  * Abdominal and pelvic CT scan, and
  * Head CT scan or MRI PET/CT fusion scan may replace scans of the chest, abdomen, and pelvis.
* Participants who have melanoma available for biopsy pre-treatment and on day 22 must consent to having those biopsies. Melanoma lesions may be in nodes, skin, soft tissue, liver, or other sites that can be accessed by core needle biopsy, or incisional or excisional biopsy, with or without image guidance.
* Participants who have had brain metastases will be eligible if all of the following are true:

  * Each brain metastasis must have been treated by surgical removal, stereotactic radiosurgery or managed to complete resolution with immunotherapy. Patients with brain lesions managed by immunotherapy without excision or radiosurgery are included provided that the brain metastases have completely resolved after systemic therapy and there are no neurologic symptoms or need for systemic therapy to control CNS-disease related symptoms.
  * There has been no evident growth of any brain metastasis since the most recent treatment. If a patient has been managed by immunotherapy alone, the prior lesions must be completely resolved.
  * No brain metastasis is > 2 cm in diameter at the time of registration
  * The most recent surgical resections or gamma-knife therapy for malignant melanoma must have been completed ≥ 1 week prior to registration.
* ECOG performance status of 0 or 1
* Ability and willingness to give informed consent
* Adequate lab function tests Age 18 years or older at registration.
* Participants must have at least two intact (undissected) axillary and/or inguinal lymph node basins

Exclusion Criteria:

* Participants who have received the following medications or treatments at any time within 4 weeks of registration:

  * Chemotherapy
  * Interferon (e.g. Intron-A®)
  * Radiation therapy (Stereotactic radiotherapy, such as gamma knife, can be used ≥ 1 week prior to registration)
  * Allergy desensitization injections
  * High doses of systemic corticosteroids, with the following qualifications and exceptions:

    * Daily doses of 10 mg predisone (or equivalent) per day administered parenterally or orally are not allowed in patients with normal adrenal and pituitary function.
    * In patients with adrenal or pituitary insufficiency replacement steroid doses are allowed.
    * Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) are permitted at low doses (less than 500 mcg fluticasone per day, or equivalent).
    * Topical and nasal corticosteroids are acceptable.
  * Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
  * Interleukins (e.g. Proleukin®)
  * Any investigational medication
  * Targeted therapies specific for mutated BRAF or for MEK
* HIV positivity or evidence of active Hepatitis C virus (testing to be done within 6 months of study entry).
* Participants who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks
* Participants who are currently receiving a checkpoint molecule blockade therapy, or who have received this therapy within the preceding 6 weeks, with the following exceptions:

  * Participants who have received a PD-1 blocking antibody (eg: pembrolizumab or nivolumab) may be enrolled 3 weeks after receiving the last dose of that antibody.
  * Participants who have been treated previously with a CTLA-4 blocking antibody either as monotherapy or as part of combination CTLA-4/PD-1 blockade will be ineligible if CTLA-4 therapy:

    1. was discontinued early for toxicity, or
    2. did not induce stable disease or objective clinical response (by RECIST or irRC criteria) lasting 6 months or more.

Note: Patients may be eligible if they have experienced progression after a period of stable disease (6 months or more) or an objective clinical response (by irRC or RECIST) (6 months or more) induced by CTLA-4 blockade or combination CTLA-4/PD-1 blockade.

Note: Similar guidelines will apply for tremelimumab or other CTLA-4 blocking antibodies.

* Participants with known or suspected allergies to any component of the vaccine.
* Participants may not have been vaccinated previously with any of the synthetic peptides included in this protocol. Participants who have received vaccinations containing agents other than the synthetic peptides included in this protocol and have recurred during or after administration of the vaccine will be eligible to enroll 12 weeks following their last vaccination.
* Pregnancy.
* Female participants must not be breastfeeding
* Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
* Participants classified according to the New York Heart Association classification as having Class III or IV heart disease.

Participants with uncontrolled diabetes, defined as having a HGB-A1C> 7.5%.

* Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

  * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring NSAID medications
  * A history of immune-related adverse events with immune therapy, if they have resolved completely.
* Participants who have another cancer diagnosis, except that the following diagnoses will be allowed:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
  * any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 2 years
* Participants with known addiction to alcohol or drugs who are actively taking those agents, or participants with recent (within 1 year) or ongoing illicit IV drug use.
* Body weight < 110 pounds at registration, due to the amount and frequency with which blood will be drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gaughan, MD, Principal Investigator — University of Virginia; Craig L. Slingluff, Jr., MD, Study Director — University of Virginia
Locations (1):
- Cancer Center at the University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened 4/29/15 Closed to enrollment December 2018. Enrollment has been slow due to changes in standard of care, especially the dominance of PD-1 blockade over CTLA-4 blockade.
  The study was closed to enrollment due to slow accrual, despite multiple revisions in the protocol to enhance enrollment.
Groups:
- 6MHP and Ipilimumab: The vaccine drug product, 6MHP, consists of 6 class II MHC-restricted peptides derived from melanoma proteins. Each vaccine consists of 200 mcg of each of the six peptides. An aqueous solution of vaccine is mixed 1/1 with Montanide ISA-51 to form water-in-oil emulsions. Vaccines are administered days 1, 8, 15, 43, 64, and 85. All peptide vaccines are administered intradermally and subcutaneously.
  Ipilimumab will be administered in accord with the official prescribing information: 3 mg/kg intravenously once every 3 weeks, for 4 doses. Ipilimumab will be administered on days 1, 22, 43, and 64.
  Ipilimumab: Checkpoint blockade inhibitor
  6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
Period: Overall Study
Arm/Group | 6MHP and Ipilimumab
Started | 3
Completed (Closed early due to slow enrollment.) | 1
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | 6MHP and Ipilimumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety (Adverse Event Profile)
Description: Adverse event profile for the combination of ipilimumab and 6MHP
Time Frame: 30 days after the last vaccination
Population: All eligible enrolled and treated patients. Partiipants analyzed for any adverse event (AE) and for dose limiting toxicities (DLT).
Measure: Count of Participants; unit: Participants
Arm/Group | 6MHP and Ipilimumab
Number analyzed (Participants) | 3
Participants
  Number of participants with DLTs | 2
  Participants with any treatment-related AEs | 3

2. Primary Outcome: CD4+ T Cell Responses in the Blood and in the Sentinel Immunized Node
Description: CD4+ T cell responses to the peptide vaccine, defined as:
  1. any CD4+ T cell response to 6 melanoma helper peptides (6MHP) in peripheral blood mononuclear cells (PBMC) with a 10 fold (or greater) increase in response over background (high response) by ex vivo ELIspot assay.
  2. CD4+ T cell high responses to 6MHP in PBMC at at least 2 consecutive time points having peripheral blood mononuclear cells (PBMC) with a 10 fold (or greater) increase in response over background by ex vivo ELIspot assay.
  3. CD4+ T cell high response to 6MHP in sentinel immunized lymph node (SIN).
Time Frame: through day 92
Measure: Count of Participants; unit: Participants
Arm/Group | 6MHP and Ipilimumab
Number analyzed (Participants) | 3
Participants
  Number with T cell response to 6MHP in PBMC | 2
  Number with T cell response at 2 consecutive times | 0
  T cell reactivity to 6MHP in SIN | 1

3. Secondary Outcome: Epitope Spreading (Epitope-spreading for CD8+ T Cells in the Blood and the Sentinel Immunized Node)
Description: An evaluation of epitope-spreading for CD8+ T cells in the blood and the sentinel immunized node that are reactive to a panel of defined melanoma antigens.
Time Frame: through day 92
Reporting Status: Not Posted, anticipated posting 2020-06

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 6MHP and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6MHP and Ipilimumab (N=3)
uveitis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6MHP and Ipilimumab (N=3)
adrenal insufficiency (Endocrine disorders) | 1 (1)
blurred vision (Eye disorders) | 1
Other (Eye disorders) | 1 — Uveitis
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Injection site reaction (General disorders) | 2 — Reaction in skin at site of vaccine administration
alanine aminotransferase increased (Investigations) | 1
aspartate aminotransferase increased (Investigations) | 1
weight loss (Investigations) | 1
anorexia (Metabolism and nutrition disorders) | 1
dehydration (Metabolism and nutrition disorders) | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1
headache (Nervous system disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
skin induration (Skin and subcutaneous tissue disorders) | 3 — Induration of skin at vaccine administration site.
skin ulceration (Skin and subcutaneous tissue disorders) | 1 — Ulceration at vaccine administration site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT02385669/Prot_SAP_000.pdf